CLINICAL TRIAL: NCT06269796
Title: Identification of Neuromotor Signs in Preschool Children Suspected of Developmental Coordination Disorder
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, George Paras, Associate Professor, University of Thessaly
Other Study IDs: little-dcdq
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Motor Skills Disorders; Child Development; Child, Preschool
Keywords: Developmental Coordination Disorder (DCD); Little Developmental Coordination Disorder Questionnaire (Little DCDQ); Bruininks-Oseretsky Test of Motor Proficiency (BOT-2); Preschool Children
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preschool Children: A prospective study was conducted, aiming at the early detection of neuromotor signs in preschool children with suspected Developmental Coordination Disorder (DCD) in Greece.The Little Developmental Coordination Disorder Questionnaire (LDCDQ) was used to evaluate motor skills of the children. Children with scores that indicated suspicion of DCD were offered the option to undergo the BOT-2 test.
  Interventions: Diagnostic Test: Little Developmental Coordination Disorder Questionnaire (LDCDQ); Diagnostic Test: Bruininks- Oseretsky Test of Motor Proficiency 2nd Edition (BOT-2)

INTERVENTIONS:
Diagnostic Test: Little Developmental Coordination Disorder Questionnaire (LDCDQ) — The Little Developmental Coordination Disorder Questionnaire (LDCDQ) is a parent questionnaire consisting of 15 items designed to screen for motor coordination difficulties in 3- and 4-year-old children. It comprises 15 items grouped into two distinct factors: gross motor skills and fine motor skills. A Likert scale is used, ranging from one to five, where one (1) indicates "Not at all like your child" and five (5) indicates "Very much like your child". The total of the 15 items is added up to obtain a total score of 75.
Diagnostic Test: Bruininks- Oseretsky Test of Motor Proficiency 2nd Edition (BOT-2) — The BOT-2 is standardized for children and adolescents aged 4 to 21 years and 11 months, and the full test takes 45 to 60 minutes to perform. The BOT-2 test was used to detect deviation from the norm and the likelihood of a diagnosis for DCD. The BOT-2 measures fine and gross motor proficiency, with subtests focusing on stability, mobility, strength, coordination, and object manipulation.

SUMMARY:
This prospective study aimed to detect neuromotor signs early in preschool children suspected of Developmental Coordination Disorder (DCD). Preschool children aged 3-5 years old from municipal kindergartens in Thessaloniki participated in this study. The Little DCDQ questionnaire and the BOT-2 (Bruininks-Oseretsky Test of Motor Proficiency) were used for assessment.

ELIGIBILITY:
Inclusion Criteria:

* Preschool children
* Aging from 3 to 5 years old

Exclusion Criteria:

* Diagnosis for medical conditions or mental retardation

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preschool children aged 3-5 from 39 municipal kindergartens in Thessaloniki, Greece, who responded to the research invitation.
Sampling Method: Non-Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Parent Screening Questionnaire for Motor Coordination Difficulties (DCD) | Complete Form - 10-15 minutes
  Little Developmental Coordination Disorder Questionnaire (LDCDQ); Unit of Measure: Likert Scale from 1 ("Not at all like your child") to 5 ("Very much like your child")
Screening Test for Detection of Developmental Coordination Disorder (DCD) | Complete Form - 45-60 minutes
  Bruininks- Oseretsky Test of Motor Proficiency 2nd Edition (BOT-2); Unit of Measure: ...

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Poulis, Prof, Study Chair — University of Thessaly
Locations (1):
- Human Performance & Rehabilitation Laboratory, Department of Physiotherapy, University of Thessaly, Lamia, Pthiotis, Greece

IPD SHARING:
Plan to Share IPD: No